CLINICAL TRIAL: NCT00662298
Title: The Pharmacokinetics and Anti-inflammatory Effects of Prednisolone in Severe Asthma
Brief Title: Prednisolone Pharmacokinetics in Severe Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2007-002084-27; REC ref number 07/H0801/119
Record Dates: First submitted 2008-04-14; First posted 2008-04-21 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: severe asthma; prednisolone pharmacokinetics; anti-inflammatory effects
MeSH Terms: conditions — Asthma | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe Asthma (Experimental)
  Interventions: Drug: prednisolone

INTERVENTIONS:
Drug: prednisolone — 40mg of prednisolone once a day for 14 days

SUMMARY:
The purpose of the study is to evaluate whether severe asthmatic subjects have abnormal prednisolone absorption, and how this might affect the anti-inflammatory effects of prednisolone.

The aims of the study are

1. to compare the effect of high dose prednisolone on clinical and physiological responses
2. to determine the effect of long-term oral prednisolone therapy on corticosteroid responsiveness and prednisolone pharmacokinetics
3. to measure the effect of high dose prednisolone for 14 days on p38 MAPK activity, GR translocation and activation of NF-kB
4. to validate an easier method of measuring corticosteroid insensitivity using whole blood, and a spot prednisolone serum level as a measure of adherence to prednisolone therapy

DETAILED DESCRIPTION:
Asthma is a disease characterized by reversible airways obstruction, bronchial hyper-responsiveness, and chronic inflammation of the bronchial mucosal lining. Currently over 5 million people (6-8% of the population) in the UK are receiving treatment for asthma. Although most patients have mild-to-moderate asthma that is well-controlled by inhaled corticosteroids (ICS), in 5-10% of asthmatics, the disease is considered severe in that symptoms and control of asthma are largely unresponsive to treatment including systemic corticosteroids (CS). This subset of patients has greater morbidity and a disproportionate need for health care support in terms of use of drugs, admissions to hospital or use of emergency services, and time off work or school. Indeed, some severe asthma patients are also on oral CS in addition to ICS, and these patients are often described as being steroid-dependent since they need oral CS in addition to ICS to maintain their asthma control. Recent studies from our laboratory have shown that patients with severe asthma have relative corticosteroid resistance as measured by the responsiveness of peripheral blood mononuclear cells and alveolar macrophages to dexamethasone.

In asthma, corticosteroid- resistance (CSR) has usually been defined on the basis of changes in baseline FEV1 (forced expiratory volume in one second) after a 14-day course of oral prednisolone of 40mg/day; an increase of less than 15% of the baseline measurement, while demonstrating a greater than 15% improvements in FEV1 following inhaled β2-agonist, has been used. Patients who showed an improvement in FEV1 of 30% or more were considered as corticosteroid-sensitive (CSS). The arbitrary cut-off response of <15% response was chosen empirically without the knowledge of the distribution of responses to oral or inhaled CS. CSR asthmatics are not completely resistant to the effects of corticosteroids, as stopping corticosteroid therapy leads to a clinical deterioration. It is not known at present whether the reduced corticosteroid responsiveness seen in severe asthma is genetically-determined or acquired, or both. Patient with CSR as defined above are not necessarily patients with severe asthma. The response of patients with severe asthma to a formal trial of oral prednisolone on lung function or inflammatory parameters has not been studied in detail. For example, it is not known whether the absorption of oral prednisolone which is commonly used to treat exacerbations of asthma is normal in patients with severe asthma. Pharmacokinetic studies have been reported in normal subjects and mild-moderate asthma, and also in CS-resistant asthmatics, and 'normal' pharmacokinetics has been reported in the latter groups. However, we need to exclude this as a potential course of relative CS-resistance in severe asthma.

Corticosteroids are known to exert anti-inflammatory effects as assessed in bronchial biopsies, which is the basis of its beneficial effects in asthma. These effects can also be assessed non-invasively using measurements of exhaled nitric oxide (eNO) or induced sputum eosinophil counts. The effect of a prednisolone trial on these measurements has not been performed. We have previously shown the value of measuring IL-8 release from whole blood as a marker of the inflammatory response. Serum IL-8 and TNF-α have been found to be higher in severe asthmatics than in the mild-moderate asthmatics. Therefore, we propose to study the response of patients with severe asthma to oral prednisolone, looking at drug levels and their anti-inflammatory effects. Anecdotally, we have found that many of our severe asthmatic patients have low prednisolone levels, even though they have been compliant with their medication. Spot levels of prednisolone (one-off measurements of blood levels) are used to check compliance. The effect of continuous oral therapy on prednisolone levels and its suppression of inflammation is unknown. It has been previously postulated that such therapy may lead to a reduction in the effectiveness of corticosteroids as an anti-inflammatory agent. Therefore, we propose to study two groups of patients with severe asthma, those on ICS alone and those on ICS plus a maintenance dose of prednisolone ranging 5-20 mg/day; the control group would be moderately-severe asthmatics who are well controlled on ICS.

The patients will be given a fourteen-day course of daily 40mg of prednisolone (non enteric-coated tablets). Subjects will attend the Asthma Lab at the Royal Brompton Hospital for screening. They will keep peak expiratory flow rate (PEFR) and symptom diary cards for 2 weeks prior to and during the two week course of prednisolone. Patients already on prednisolone will have the maintenance dose increased to 40mg. There will be 5 study visits.

On Visits 2 and 4, patients will be fasting overnight and will have the blood tests at time 0 hours. They will then take the prednisolone with or after having their breakfast. Sputum and blood samples will be taken, spirometry and exhaled nitric oxide measured at various time intervals as specified in the protocol. Visits 3 and 5 will be 24 hours post 1st and last prednisolone dose

ELIGIBILITY:
Inclusion Criteria:

* for severe asthmatics:

  * Physician diagnosis of asthma
  * Aged 18 - 70
  * Non-smokers or ex-smokers with less than 5 pack/year history
  * Major characteristics (at least one of the following criteria)
  * Treatment with continuous or near continuous (>50% of year) oral corticosteroids
  * Requirement for treatment with high dose inhaled corticosteroids (ICS)
  * Minor characteristics (at least 2 out of the following)

    1. Requirement for daily treatment with a controller medication in addition to ICS e.g. LABA, theophylline, leukotriene antagonist
    2. Asthma symptoms requiring SABA on a daily or near daily basis
    3. Persistent airways obstruction (FEV1 <80% predicted, diurnal PEF variation >20%)
    4. One or more emergency care visits for asthma per year
    5. 3 or more steroid "bursts" per year
    6. Prompt deterioration with ≤ 25% reduction in oral or ICS
    7. Near fatal asthma event in the past
* for moderately-severe asthma:

  * Physician diagnosis of asthma
  * Aged 18 - 70
  * Non-smokers or ex-smokers with less than 5 pack/year history
  * Less than 2 courses of prednisolone per year
  * Taking up to 2000 mcg of inhaled corticosteroid (BDP equivalent) per day
  * Stable asthma for at least 6 months prior to enrollment

Exclusion Criteria:

* Current smokers, or less than 3 years since quitting smoking
* Less than 4 weeks from an exacerbation
* Diabetes
* Active peptic ulceration
* Previous history of psychiatric disturbances on high dose prednisolone
* On steroid-sparing agent or immunosuppressant such as azathioprine, methotrexate and ciclosporin
* Concomitant anti-IgE therapy
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian F Chung, Principal Investigator — Imperial College London
Locations (1):
- Asthma Laboratory, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severe Asthma
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Severe Asthma
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Serum Prednisolone Levels Over 24 Hours
Time Frame: 2h, 6h, 24h
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Severe Asthma
Number analyzed (Participants) | 5
nmol/l
  2h | 800 (600)
  6h | 700 (500)
  24h | NA (NA) — NA (Not Available), below level of detection

2. Primary Outcome: Change in FEV1 24 Hours Post Prednisolone
Time Frame: 14 days
Population: No data collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

3. Primary Outcome: Changes in eNO, Sputum Eosinophils and Inflammatory Mediators Over 24 Hours
Time Frame: 14 days
Population: Data not collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

4. Secondary Outcome: Difference Between Baseline and Day 14 in Serum Prednisolone Levels
Time Frame: Baseline, 14 days
Measure: Mean (Full Range); unit: nmol/litres
Arm/Group | Severe Asthma
Number analyzed (Participants) | 5
nmol/litres
  baseline | 2.0 [1.45 to 2.73]
  14days | 2.11 [1.61 to 2.82]

5. Secondary Outcome: Difference in FEV1 Between Day 1 and Day 14
Time Frame: 14 days
Population: Data were not collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

6. Secondary Outcome: Difference in Inflammatory Markers Between Day 1 and Day 14
Time Frame: 14 days
Population: Data were not collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in Asthma Control Symptoms Before and After Treatment
Time Frame: 14 days
Population: Data were not collected.
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Severe Asthma
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes